CLINICAL TRIAL: NCT02444260
Title: Improving Patient Outcomes With Inguinal Hernioplasty - a Randomized Controlled Trial of Local Anaesthesia Versus Local Anaesthesia and Conscious Sedation
Brief Title: A Trial of Local Anaesthesia Versus Local Anaesthesia and Conscious Sedation for Hernioplasty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECP342,12/13
Record Dates: First submitted 2015-04-28; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-03

CONDITIONS: Inguinal Hernia; Anesthesia, Local; Conscious Sedation
Keywords: Inguinal Hernia,; Local Anesthesia; Randomized Clinical trial; HERNIOPLASTY
MeSH Terms: conditions — Hernia, Inguinal | interventions — Midazolam; Sodium Chloride; Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Normal Saline (Sham Comparator): Intravenous Normal Saline plus Lignocaine HCl (1%) - administered by wound infiltration to a maximum dose of 4.5mg/kg ; Bupivocaine HCl (0.25%) - administered by wound infiltration to a maximum dose of 2 mg/kg plus i
  Interventions: Drug: Intravenous Normal Saline; Drug: Bupivocaine; Drug: Lignocaine HCl
- Midazolam (Active Comparator): Lignocaine HCl (1%) - administered by wound infiltration to a maximum dose of 4.5mg/kg Bupivocaine HCl (0.25%) - administered by wound infiltration to a maximum dose of 2 mg/kg plus Midazolam - administered intravenously. 1 mg given stat. Titrated by 1 mg to a maximum dose of 10 mg.
  Interventions: Drug: Midazolam; Drug: Bupivocaine; Drug: Lignocaine HCl

INTERVENTIONS:
Drug: Midazolam — Midazolam will administered intravenously. 1 mg given stat. Titrated by 1 mg to a maximum dose of 10 mg. Additional sedation will be given to achieve and maintain a score of 2-3 on the Ramsay sedation scale during the procedure, up to the maximum dose of 10mg.
  Other Names: Dormicum
  Arms: Midazolam
Drug: Intravenous Normal Saline — Intravenous normal saline will be infused by non-blinded anaesthetist
  Other Names: 0.9% sodium chloride solution
  Arms: Intravenous Normal Saline
Drug: Bupivocaine — Bupivcaine 0.25% solution administered by wound infiltration to a maximum dose of 2 mg/kg
  Other Names: Marcaine
Drug: Lignocaine HCl — Lignocaine !% solution administered by wound infiltration to a maximum dose of 4.5mg/kg
  Other Names: xylocaine

SUMMARY:
The aim of this RCT is to compare patient outcomes of inguinal hernioplasty under Local Anaesthesia alone versus Local Anaesthesia and Conscious Sedation

Specific study objectives are to determine the effect of conscious sedation on:

(i) patient satisfaction (ii) postoperative pain (iii) time to discharge (iv) intraoperative complications (v) postoperative functional status (vi) short-term postoperative complications (vii) long-term postoperative complications

ELIGIBILITY:
Inclusion Criteria:

* Reducible inguinal hernia

Exclusion Criteria:

* Renal, hepatic, respiratory, cardiovascular, neurologic or psychiatric disease
* Body mass index < 18.5 kg/m2 or > 30 kg/m2
* Recurrent inguinal hernias
* Bilateral inguinal hernias
* Large inguinoscrotal hernias
* Incarcerated hernia
* Allergies to local anaesthetic and sedative agents
* Pregnancy
* Lactation
* Chronic pain syndromes
* Anxiety disorders
* Marijuana use
* Long term use of opioid or sedative agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction as assessed with the Iowa Satisfaction with Anesthesia Scale | 1 year
  Change in the Iowa Satisfaction with Anesthesia Scale from baseline (pre-discharge assessment)

SECONDARY OUTCOMES:
Operative time | 2 weeks
Frequency (total count) of postoperative complications using a questionaire | 1 year
Post-operative assessment of physical activity using Activities Assessment Scale | 1 year
Time to discharge | 2 weeks
change in postoperative pain score from baseline assessed with visual analog scale | 1 year
  change in postoperative pain from baseline (pre-discharge assessment) assessed with visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of the West Indies, mona, Kingston, Please Select, Jamaica

REFERENCES:
- [Derived] Leake PA, Toppin PJ, Reid M, Plummer JM, Roberts PO, Harding-Goldson H, McFarlane ME. Local Anesthesia Versus Local Anesthesia and Conscious Sedation for Inguinal Hernioplasty: Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2017 Feb 7;6(2):e20. doi: 10.2196/resprot.6754. PMID 28174148